CLINICAL TRIAL: NCT05275426
Title: A Phase II Study of Oral CHK1 Inhibitor LY2880070 in Combination With Low-Dose Gemcitabine in Patients With Relapsed or Refractory Ewing Sarcoma, Ewing-like Sarcoma, and Desmoplastic Small Round Cell Tumor
Brief Title: A Study of LY2880070 and Gemcitabine in People With Ewing Sarcoma,Ewing-Like Sarcoma, and Desmoplastic Small Round Cell Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-428
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Ewing Sarcoma; Ewing-Like Sarcoma
Keywords: Ewing Sarcoma; Ewing-Like Sarcoma; LY2880070; Gemcitabine; 21-428; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ewing sarcoma (Experimental): Participants have a diagnosis of Ewing sarcoma as molecularly defined by an EWSR1 fusion with an ETS-transcription factor family member including FLI1, ERG, ETV1, ETV4, and FEV
  Interventions: Drug: LY2880070; Drug: Gemcitabine

INTERVENTIONS:
Drug: LY2880070 — Patients will receive treatment in 21-day cycles with LY2880070 50 mg twice daily orally on days 2-6, 9-13, and 16-20
Drug: Gemcitabine — Participants will receive treatment in 21-day cycles with gemcitabine 100 mg/m2 intravenously on days 1, 8 and optionally on day 15

SUMMARY:
The purpose of this study is to find out whether LY2880070 combined with the chemotherapy drug gemcitabine is an effective treatment for Ewing sarcoma or Ewing-like sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Consent/Assent: all patients and/or their parents or legally authorized representatives must sign written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Weight/Age: patients must be ≥40 kg at the time of study enrollment, but may be of any age
* Diagnosis: Patients must have histologically documented locally advanced or metastatic disease confirmed at MSK as follows:

  * Main cohort: Ewing sarcoma as molecularly defined by an EWSR1 fusion with an ETS-transcription factor family member including FLI1, ERG, ETV1, ETV4, and FEV
  * Pilot cohort: Ewing-like sarcomas including CIC-rearranged sarcoma, BCOR-rearranged sarcoma, and sarcomas with a rearrangement between EWSR1 and a non-ETS family gene or desmoplastic small round cell tumor as molecularly defined by an EWSR1-WT1 fusion

Note: Any patient being enrolled into the pilot cohort that does not have a CIC, BCOR- rearranged sarcoma, or desmoplastic small round cell tumor will be reviewed with study pathologist, Dr. Cristina Antonescu, to ensure the categorization as Ewing-like sarcoma is appropriate

* Patients must be able to swallow capsules
* Therapeutic options: patient's current disease state must be one which has failed standard cytotoxic chemotherapy including cyclophosphamide/doxorubicin/vincristine and ifosfamide/etoposide
* Disease Status: patients must have measurable disease based on RECIST 1.1
* Performance level: Karnofsky ≥70% for patients >16 years of age and Lansky ≥70 for patients ≤16 years of age
* Prior Therapy: patients may have had any number of regimens and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment

Note: Patients who have previously received gemcitabine will be allowed unless they had hypersensitivity or unacceptable toxicity attributed to gemcitabine

* ≥ 21 days must have elapsed after the last dose of cytotoxic or myelosuppressive chemotherapy and patients must have recovered from the acute toxic effects of these agents (other than alopecia)
* ≥ 14 days must have elapsed after radiation therapy, and toxicity related to prior radiation therapy must be recovered to grade ≤ 1
* ≥ 21 days must have elapsed after the last dose of antibody therapy, and toxicity related to prior antibody therapy must be recovered to grade ≤ 1

Organ Function Requirements:

* Adequate bone marrow function defined as:

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hemoglobin ≥ 8 g/dl
* Adequate renal function defined as estimated glomerular filtration (eGFR) rate ≥ 60 mL/min/1.73m2:

  * as estimated by CKD-EPI equation for patients ≥ 18 years of age OR
  * As estimated by cystatin C for patients < 18 years of age
* Adequate liver function defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal for age
  * AST or ALT ≤ 2.5 x upper limit of normal for patients without liver metastases
  * AST or ALT ≤ 5 x upper limit of normal for patients with liver metastases
  * Serum albumin ≥ 2.5 g/dl
* Adequate cardiac function defined as:

  * Left ventricular ejection fraction (LVEF) >45% as measured on echocardiogram, cardiac MRI, or MUGA
  * QTc < 470 ms on screening 12 lead electrocardiogram
* Pregnancy/Contraception

  * Post-menarchal females must have a negative urine or serum pregnancy test at screening and ≤ 24 hours prior to study treatment
  * Males or females of reproductive potential must be willing to use a barrier method of contraception throughout the course of the study and for 6 months after completing study treatment

Exclusion Criteria:

* Patients for whom the investigator deems that gemcitabine is not appropriate
* Patients who have an uncontrolled infection
* Central Nervous System (CNS) Metastases

  * Patients who have symptomatic central nervous system (CNS) metastases. Note: patients with treated and asymptomatic CNS metastases are eligible.
  * Patients with CNS metastases requiring corticosteroids for management
  * If the treatment of CNS disease requires anticonvulsants, the dose must have been stable for ≥ 4 weeks.
* Patients who are pregnant or breast feeding
* Patients who have a history of Torsades de Pointes, carry a diagnosis of congestive heart failure, or have a family history of prolonged QT syndrome
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Patients with known hypersensitivity to gemcitabine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Best overall response rate | 6 months
  The ORR will include complete response and partial response (CR+PR) as defined using RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org